CLINICAL TRIAL: NCT03468465
Title: Peripheral Transcutaneous Neuromodulation of the Post-tibial Nerve (T-PTNS) for Solifenacin 10 mg. in the Treatment of Hyperactive Bladder Syndrome: no Inferiority Phase IV Randomized Clinical Trial
Brief Title: Peripheral Transcutaneous Neuromodulation of the Post-tibial Nerve for Solifenacin 10 mg. Hyperactive Bladder Syndrome
Acronym: SOLITENS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FFIS/2017/01/SLT; 2017-000605-20 (EudraCT Number)
Record Dates: First submitted 2018-02-20; First posted 2018-03-16 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Urinary Incontinence
Keywords: Hyperactive Bladder Syndrome
MeSH Terms: conditions — Urinary Incontinence | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical device: Transcutaneous electrical neurostimulation (Experimental): Medical device 4 weeks with daily sessions of 30 minutes
  Interventions: Device: Neuro-Muscular Stimulators (NMS)
- Solifenacin (Active Comparator): 10 mg tablet daily during 75 days maximum
  Interventions: Drug: Solifenacin Succinate

INTERVENTIONS:
Drug: Solifenacin Succinate — 10 mg tablet daily during 75 days maximum
  Other Names: Vesicare
  Arms: Solifenacin
Device: Neuro-Muscular Stimulators (NMS) — Treatment with T-PTNS will include a first induction period of 4 weeks with daily sessions of 30 minutes duration and performed at each subject's home (Monday through Friday, resting weekends) and a second recall period of 2 additional months, with a session every 4 weeks that will be held at the healthcare center. In total there will be 20 sessions in the induction period and 2 in the recall period
  Other Names: T-PTNS
  Arms: Medical device: Transcutaneous electrical neurostimulation

SUMMARY:
* To determine if the T-PTNS is not inferior in the short term (3 months) to one of the usual pharmacological treatments (Solifenacin) in the treatment of hyperactive bladder syndrome and with respect to the percentage of patients that improve 50% any of the 3 signs (Urinary frequency, diurnal / nocturnal frequency, urgency and urinary incontinence).
* To determine prognostic factors associated with insufficient improvement (less than 50% in the 3 main signs of hyperactive bladder syndrome (urinary frequency, urgency and urinary incontinence frequency) after treatment with T-PTNS and Solifenacin.

DETAILED DESCRIPTION:
Patients will be randomized to receive the usual standard treatment with Solifenacin or treatment based on peripheral unilateral transcutaneous neuromodulation of the posterior tibial nerve .

ELIGIBILITY:
Inclusion Criteria:

* Women> 18 years, diagnosed with hyperactive bladder syndrome for at least 6 months of evolution and who have taken Beta 3 agonists

Exclusion Criteria:

* Patients who can contribute biased information: have previously consumed and abandoned anticholinergic drugs due to lack of efficacy or side effects; Suffering from hyperactive bladder of neurogenic origin (multiple sclerosis, Parkinson's, spinal cord injury); Present cystocele or any pelvic organ prolapse> 2 according to Pelvic Organ Prolapse-Q classification
* Patients who may become worse with the interventions envisaged in the study: being a implantable automatic defibrillators; With cutaneous alterations in lower extremities that prevent the placement of electrodes on the surface; Women who are pregnant or who may be pregnant during the duration of the clinical trial (prior and at each evaluation visit urine Bhcg will be requested to rule out pregnancy) or patients who are not able to manage transcutaneous electrical neurostimulation on an outpatient basis ) Or patients in whom Solifenacin is contraindicated: urinary retention, severe gastrointestinal disorders (including toxic megacolon), myasthenia gravis, or narrow-angle glaucoma, and in patients at risk of these conditions as hypersensitive at first Active or to any of the excipients, undergoing hemodialysis, with moderate hepatic insufficiency or severe renal insufficiency or in simultaneous treatment with a potent inhibitor of CYP3A4, eg ketoconazole.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate whether treatment with T-PTNS is not less than 3 months compared to the current standard pharmacological treatments regarding the episodes of urgency, urinary frequency, incontinence and nocturia, all measured with the 3-day voiding diary | 12 weeks
  3- day voiding diary

CONTACTS AND LOCATIONS:
Overall Officials: José David Jiménez Parra, MD, Principal Investigator — Hospital Rafael Méndez (Lorca, Murcia. SPAIN); María Luisa María Luisa, MD, Principal Investigator — Hospital Clínica Universitario Virgen de la Arrixaca (SPAIN); José Felix Escudero Bregante, MD, Principal Investigator — Hospital Clínico Universitario Virgen de la Arrixaca (SPAIN); Julián Oñate, MD, Principal Investigator — Hospital General Universitario Reina Sofía (SPAIN); Ana Isabel López López, MD, Principal Investigator — Hospital Clínico Universitario San Juan (SPAIN)
Locations (1):
- Hospital Clínico Universtario Virgen de la Arrixaca, El Palmar, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No